CLINICAL TRIAL: NCT02688582
Title: A Study to Evaluate the Predictive Performance of a Target-controlled Infusion Model for the Administration of Cefepime to Intensive Care Patients
Brief Title: Target-controlled Infusion Model for Cefepime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: University Ghent (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Stijn Jonckheere, Principal Investigator, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/005
Record Dates: First submitted 2016-02-06; First posted 2016-02-23 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Antimicrobial Treatment
Keywords: Target Controlled Infusion; Pharmacokinetics; Cefepime; critically ill patients

ARMS (1):
- TCI group (Experimental): Patients who receive cefepime based on TCI for a maximum of 5 days with a target concentration of cefepime of 16 mg/L.
  Interventions: Other: TCI group

INTERVENTIONS:
Other: TCI group — Drug: cefepime, Device: Target Controlled Infusion pump connected to Rugloop vII software

SUMMARY:
For this study, a previously developed population pharmacokinetic (popPK) model for cefepime (Jonckheere et al., submitted to JAC) was programmed in Rugloop vII, which is a software program to drive an infusion pump. By entering patient data (such as gender, serum creatinine, age and weight) in Rugloop II, a patient-specific dose will be calculated and given to the patient. This concept is known as Target Controlled Infusion (TCI). The aim of this study is to prospectively validate the popPK model using TCI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 years of age or older, admitted to the hospital ICU and requiring administration of cefepime as part of their treatment
* Patients within the weight range of 50 -120kg
* Patients with calculated creatinine clearance within the range 15 to > 90 ml/min, allocated to one of three groups as described above.
* Written informed consent, or if not possible surrogate consent, or if not possible declaration for inclusion in an emergency, patient informed consent being signed as soon as possible.
* Patient with an arterial catheter in place for other reason than the current study purpose

Exclusion Criteria:

* Patients displaying acute or chronic renal failure requiring renal replacement therapy
* Pregnancy
* Moribund patients
* Known sensitivity or allergy to cefepime
* Inclusion in another study involving antimicrobial treatment.
* Patient participating in a research for which a period of exclusion is currently required by other study protocol, ethical committee or health authority.
* Patient already previously included in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Median Absolute Preditive Error (MdAPE, %) of predicted versus measured cefepime plasma concentrations (mg/L) | During the first 5 days of cefepime therapy

SECONDARY OUTCOMES:
Percentage of patients with Neurotoxicity related to cefepime based on Naranjo criteria | Evaluation during the first 5 days of cefepime therapy
Negativation of microbiological cultures | Evaluation during the first 5 days of cefepime therapy
  When applicable, evaluation of semi-quantitative culture of clinical samples (e.g. respiratory samples). This is not mandatory for study inclusion.
Percentage of patients with clinical cure | At the end of the study (maximum 5 days after inclusion)
  Clinical cure when all criteria are met:
  * Patient not deceased
  * WBC count between 4000/µL and 11000/µL OR decreased by 25% relative to peak value
  * CRP decrease of 50% relative to peak value
  * If respiratory infection: i) absence or decrease in sputa/tracheal secretions; ii) extubated and not re-intubated within 24h after cessation of cefepime (if relevant)
  * Body temperature between 35°C and 38°C

REFERENCES:
- [Derived] Jonckheere S, De Neve N, Verbeke J, De Decker K, Brandt I, Boel A, Van Bocxlaer J, Struys MMRF, Colin PJ. Target-Controlled Infusion of Cefepime in Critically Ill Patients. Antimicrob Agents Chemother. 2019 Dec 20;64(1):e01552-19. doi: 10.1128/AAC.01552-19. Print 2019 Dec 20. PMID 31685467